CLINICAL TRIAL: NCT05816083
Title: Development and Evaluation of a Virtual Reality Tool for At-Risk Trauma-Exposed Young People
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105369
Record Dates: First submitted 2023-02-23; First posted 2023-04-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorders; HIV Infections
Keywords: substance use disorders; alcohol use; substance use; HIV infections; HIV risk; virtual reality
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality (Experimental): All participants will receive the same intervention
  Interventions: Behavioral: Virtual Reality Tool

INTERVENTIONS:
Behavioral: Virtual Reality Tool — Virtual Reality Tool for At-Risk Trauma-Exposed Young People

SUMMARY:
This is a multi-phased study, funded through a National Institute on Drug Abuse (NIDA) K24 grant that aims to ultimately refine a virtual reality tool through qualitative and quantitative research targeting HIV and substance abuse risk behavior among at-risk young people who have experienced psychosocial trauma. Participants eligible for this study include young men who have sex with men (YMSM)/individuals who are romantically/physically attracted to men and adolescents with substance use disorder (SUD) between the ages of 15 - 30 and have experienced at least one traumatic event in their lifetime. Frontline healthcare workers who work within these populations are eligible for the study as well.

DETAILED DESCRIPTION:
YMSM and adolescents with SUD participants will complete 3 study sessions. During session 1, informed consent and baseline measures are administered. Approximately one week later, during session 2, participants use and assess the virtual reality tool. Approximately one week later, during session 3, baseline assessments are re-administered.

ELIGIBILITY:
Inclusion Criteria for YMSM are as follows:

* Someone who identifies as a YMSM or identifies as someone with romantic or physical attraction to individuals who identify as men
* Is aged 15-30 years
* Have experienced at least one ITE in lifetime (i.e., sexual assault, physical assault, witnessed domestic or community violence)
* Report being consensually sexually active or planning to become sexually active with a partner in the next 12 months
* Live in the Charleston, SC/Tri-county area

Inclusion Criteria for adolescents with SUD are as follows:

* Someone who reports using substances in the past year (for participants ages 15-17) or the past 6 months (for participants ages 18-30)
* Is aged 15-30 years
* Have experienced at least one ITE in lifetime (i.e., sexual assault, physical assault, witnessed domestic or community violence)
* Report being consensually sexually active or planning to become sexually active with a partner in the next 12 months
* Live in the Charleston, SC/Tri-county area

Inclusion Criteria for front line healthcare workers are as follows:

* works directly with adolescents who have experienced ITE and/or
* works directly with adolescents or young adults with SUD and/or
* works directly with YMSM and/or
* works directly with and/or adolescent or young adults who are HIV-positive

Exclusion Criteria for all participants are as follows:

* exhibits psychotic symptoms;
* exhibits significant cognitive disability;
* reports a history of Pervasive Developmental Disorder;
* has active suicidal or homicidal ideations
* self-reports high levels of motion sickness

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Quantity and Frequency of Substance Use | Day 0 (Session 1) up to Day 14 (Session 3)
  The Timeline Follow Back (TLFB) is a validated, subjective measure that uses a calendar for people to provide estimates of substance use (drugs/alcohol) on a daily basis, retrospectively. Key dates and calendars are used to aid in memory recall. The measure is beneficial in both clinical and research environments. Over time, the TLFB looks for a decrease in substance use. Higher numbers of substance use are indicative of greater substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Danielson, Principal Investigator — Medical University of South Carolina
Locations (1):
- National Crime Victims Research and Treatment Center, Charleston, South Carolina, United States